CLINICAL TRIAL: NCT03893487
Title: A Target Validation Study of Fimepinostat in Children and Young Adults With Newly Diagnosed Diffuse Intrinsic Pontine Glioma (DIPG), Recurrent Medulloblastoma, or Recurrent High-Grade Glioma (HGG)
Brief Title: Fimepinostat in Treating Brain Tumors in Children and Young Adults
Acronym: PNOC016
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sabine Mueller, MD, PhD (Other)
Collaborators: Pediatric Neuro-Oncology Consortium (Other); Cannonball Kids' Cancer Foundation (Other); Curis, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Sabine Mueller, MD, PhD, Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18086; NCI-2019-00144 (Other: NCI Clinical Trials Reporting Program (CTRP)); PNOC016 (Other: Pediatric Neuro-Oncology Consortium)
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Diffuse Intrinsic Pontine Glioma; Recurrent Anaplastic Astrocytoma; Recurrent Glioblastoma; Recurrent Malignant Glioma; Recurrent Medulloblastoma
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Astrocytoma; Glioblastoma; Glioma; Medulloblastoma | interventions — fimepinostat; CUDC-907

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (fimepinostat, tumor resection) (Experimental): Patients receive fimepinostat by mouth once daily, on Days -2 to 0. Within 2 hours of receiving fimepinostat on Day 0, patients undergo tumor resection or biopsy as part of their standard of care.
  MAINTENANCE PHASE: Patients receive fimepinostat by mouth, once daily for days 1-5 each week. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity for up to 12 months from the time treatment begins. Should patients continue to derive clinical benefit, and not experience excess toxicity or progression, patients can continue to receive drug for up to 24 months or longer pending discussion with study chairs and study sponsor.
  Interventions: Drug: Fimepinostat; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Fimepinostat — Fimepinostat capsules
  Other Names: CUDC-907
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This trial studies how well fimepinostat works in treating patients with newly diagnosed diffuse intrinsic pontine glioma, or medulloblastoma, or high-grade glioma that have come back. Fimepinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To confirm penetration of fimepinostat across the blood brain barrier (BBB) in children and young adults with newly diagnosed diffuse intrinsic pontine glioma (DIPG), recurrent medulloblastoma, or recurrent high-grade glioma (HGG) by measuring concentration of fimepinostat and metabolite in primary tumor tissue.

EXPLORATORY OBJECTIVES:

I. To assess pharmacokinetics (PK) of fimepinostat in plasma and tumor tissue of children and young adults with newly diagnosed DIPG, recurrent medulloblastoma, or recurrent HGG.

II. To assess pharmacodynamics (PD) of fimepinostat in children and young adults with newly diagnosed DIPG, recurrent medulloblastoma, or recurrent HGG as measured by phosphorylation and acetylation in tumor tissue.

III. To correlate acetylation and phosphorylation in tumor tissue with tissue and plasma PK levels.

IV. To assess the safety and tolerability of fimepinostat in children and young adults with newly diagnosed DIPG, recurrent medulloblastoma, or recurrent HGG.

V. To assess preliminary efficacy of fimepinostat given as monotherapy after surgery in children and young adults with newly diagnosed DIPG, recurrent medulloblastoma, or recurrent HGG, as based on progression-free survival (PFS) and objective response rate (ORR) as appropriate.

OUTLINE:

Patients receive fimepinostat orally (PO) once daily (QD) on days -2 to 0. Within 2 hours of receiving fimepinostat on day 0, patients undergo tumor resection.

MAINTENANCE PHASE: Patients receive fimepinostat by mouth, once daily for days 1-5 each week. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity for up to 12 months from the time treatment begins. Should patients continue to derive clinical benefit, and not experience excess toxicity or progression, patients can continue to receive drug for up to 24 months or longer pending discussion with study chairs and study sponsor.

After completion of study treatment, patients are followed up at 30 days, then every 3 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have one of the following histologically confirmed diagnoses (histologic confirmation from initial diagnosis acceptable, as appropriate):

  * Stratum A: Newly diagnosed diffuse intrinsic pontine glioma (WHO grade II-IV) - this stratum does not require tissue confirmation at time of enrollment, but diagnostic confirmation will be required to continue on study after biopsy. Patients with newly diagnosed DIPG will be eligible to enroll before or after standard of care radiation, but must be eligible for a biopsy. Newly diagnosed DIPG stratum should not have received prior therapy before the initiation of fimepinostat, with the exception of those patients who received temozolomide during radiation therapy or who previously received radiation as per standard of care and have not yet undergone a biopsy. All patients who have received therapy other than radiation and temozolomide should be discussed with study chair(s) prior to enrollment. Patients enrolling after standard of care radiation must be enrolled within 14 weeks of completion of radiotherapy.
  * Stratum B: Recurrent medulloblastoma (WHO grade IV), any molecular subtype
  * Stratum C: Recurrent high-grade glioma (HGG), including anaplastic astrocytoma (WHO grade III) and glioblastoma (WHO grade IV)

    * Stratum B & C: Patients in the recurrent medulloblastoma or recurrent HGG arm can have locally recurrent or disseminated disease, provided resection/biopsy would still be clinically indicated. Disseminated disease can be diagnosed by imaging or Cerebrospinal fluid (CSF) cytology. Recurrent DIPG will be eligible for stratum C; however, eligibility requires biopsy/resection is feasible in a region of tumor outside of the pons (i.e. cerebellar extension or new metastatic site). These patients should be discussed with study chair(s) prior to enrollment
* Patients must be able to swallow intact fimepinostat capsules or mini-tabs without chewing or crushing
* Patients must have body surface area (BSA) >= 0.5 m^2
* Patients must undergo tumor tissue collection as part of their standard of care

  * Minimum possible tissue collected must be equivalent to about 4-6 stereotactic core biopsies
* Prior Therapy: Patients in the medulloblastoma and HGG strata will be allowed to have undergone prior therapy including surgery, chemotherapy, and radiation therapy. Patients in the newly diagnosed DIPG stratum should not have received prior therapy before the initiation of fimepinostat, with the exception of those patients who received temozolomide during radiation therapy or who previously received radiation as per standard of care and have not yet undergone a biopsy. All patients who have received therapy other than radiation and temozolomide should be discussed with study chair(s) prior to enrollment. Patients must have fully recovered from acute side effects related to previous anti-cancer therapies. Patients undergoing radiation during protocol therapy will not be permitted to receive other concomitant agents with radiation and pending initiation of maintenance with fimepinostat

  * Myelosuppressive chemotherapy: At least 21 days after last dose of myelosuppressive chemotherapy (42 days if prior nitrosourea)
  * Hematopoietic growth factors: At least 14 days after last dose of a long-acting growth factor or 7 days after short-acting growth factor or beyond time during which adverse events are known to occur
  * Biologic (anti-neoplastic agent): At least 7 days after last dose of a biologic agent or beyond time during which adverse events are known to occur
  * Monoclonal antibodies: At least 21 days after last dose of monoclonal antibody
  * Radiotherapy:

    * At least 2 weeks after local palliative radiotherapy (XRT)
    * At least 3 months from craniospinal XRT, or XRT to > 50% pelvis
  * Surgery:

    * At least 21 days from major surgery (biopsy and central line placement/removal are not considered major)
* Corticosteroids: Subjects who are receiving dexamethasone must be on a stable or decreasing dose for at least 7 days prior to enrollment
* Peripheral absolute neutrophil count (ANC) >= 1000/mm^3
* Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 milliliters (mL)/minute (min)/1.73 m^2 or
* A serum creatinine based on age/gender as follows:

  * Age: Maximum Serum Creatinine (mg/dL)
  * 3 to < 6 years: 0.8 (male), 0.8 (female)
  * 6 to < 10 years: 1 (male), 1 (female)
  * 10 to < 13 years: 1.2 (male), 1.2 (female)
  * 13 to < 16 years: 1.5 (male), 1.4 (female)
  * >= 16 years: 1.7 (male), 1.4 (female)
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT)/alanine aminotransferase (ALT) =< 110 U/L
* Serum albumin >= 2 g/dL
* Neurologic function:

  * Subjects with seizure disorder may be enrolled if well controlled
* Gastrointestinal function:

  * Diarrhea < grade 2 by Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0
* Metabolic function:

  * Non-fasting glucose < 125 mg/dL without the use of antihyperglycemic agents

    * If non-fasting glucose > 125 mg/dL, a fasting glucose should be done. If fasting glucose =< 160 mg/dL without the use of antihyperglycemic agents, patient will meet adequate metabolic function criteria
* Cardiac function: corrected QT (QTc) < 480 msec
* The effects of fimepinostat on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and 30 days after completion of fimepinostat administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* A legal parent/guardian or patient must be able to understand, and willing to sign, a written informed consent and assent document, as appropriate

Exclusion Criteria:

* Subjects who have not recovered from acute adverse events due to therapeutic agents administered more than 4 weeks earlier
* Patients must not have received prior therapy with single-agent or combination histone deacetylase (HDAC) and Phosphatidylinositol-4,5-bisphosphate 3-kinase (PI3K) inhibitors
* Subjects who are receiving any other investigational agent
* History of allergic reaction to compounds of similar chemical or biological composition to fimepinostat
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements
* Patients with active human immunodeficiency virus (HIV) infection and with potential life-threatening consequences associated with immune-suppressive therapy
* Patients with history of type 1 or 2 diabetes mellitus
* Patients with gastrointestinal condition that could interfere with absorption or metabolism of fimepinostat

Ages: 3 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Penetration of fimepinostat across the blood brain barrier (BBB) | During surgery or biopsy
  Will be analyzed using descriptive statistics from results of fimepinostat concentrations measured within the tumor tissue collected at the time of a standard of care surgery or biopsy. Within each strata, Simon's two-stage design will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Mueller, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (19):
- United States (18):
  - Children's Hospital Los Angeles (CHLA), Los Angeles, California
  - Rady Children's Hospital, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Children's Minnesota Research Institute, Minneapolis, Minnesota
  - Washington University in St Louis, St Louis, Missouri
  - Nationwide Children's, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - University of Utah, Children's Primary, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- The University Children's Hospital in Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data after de-identification
Supporting Information: Study Protocol